CLINICAL TRIAL: NCT00056654
Title: Pharmacokinetic, Safety and Efficacy Study of a Six-Month Depot Formulation of Leuprolide in Subjects With Prostatic Carcinoma
Brief Title: Study of a 6-Month Sustained-Release Formulation of Leuprolide Acetate in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Peter Bacher, Global Project Head, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C02-008
Record Dates: First submitted 2003-03-20; First posted 2003-03-21 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-09

CONDITIONS: Prostatic Neoplasms
Keywords: Leuprolide; Prostatic Neoplasms; Testosterone; Prostate-specific Antigen; Pharmacokinetics; luprolide acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Leuprolide acetate

INTERVENTIONS:
Drug: Leuprolide acetate — 45 mg Intramuscular injection 6 month depot formulation

SUMMARY:
The primary purpose of the study is to determine if a new sustained-release 45 mg (depot) formulation of leuprolide acetate will reduce serum testosterone levels to and maintain them at medically castrate levels in subjects with prostatic adenocarcinoma.

DETAILED DESCRIPTION:
The primary purpose of the study is to determine if a new sustained-release 45 mg (depot) formulation of leuprolide acetate administered once every 26 weeks for 1 year, will lower testosterone levels to and maintain them at medically castrate levels in subjects with prostatic adenocarcinoma. This study will also evaluate the pharmacokinetic profile of the 45 mg formulation and assess the safety of this formulation.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of prostate cancer
* Need for androgen deprivation treatment for 1 year
* Serum testosterone level ≥ 150 ng/dL
* Life expectancy of at least 18 months
* ECOG Performance status grades 0,1 or 2

Exclusion Criteria:

* Hypersensitivity to leuprolide acetate or polylactic acid
* History of bilateral orchiectomy, adrenalectomy, or hypophysectomy
* History of hypogonadism

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2003-03; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Suppression of serum testosterone (<=50 ng/dL) and maintenance of serum testosterone suppression once suppression is achieved for individual subjects. | Day 32 through Week 52

SECONDARY OUTCOMES:
Change from baseline in Eastern Cooperative Oncology Group (ECOG) performance status. | Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and Final Visit
Change from baseline in symptom severity (bone pain, pain on urination, urination difficulty). | Weeks 1, 4, 8, 12, 16, 20, 24, 26, 27, 28, 30, 32, 36, 40, 44, 48, 52 and Final Visit
Change from baseline in prostate specific antigen (PSA). | Weeks 1, 12, 26, 27, 30, 40, 52 and Final Visit
Change from baseline in prostatic acid phosphatase (PAP). | Weeks 1, 12, 26, 40, 52 and Final Visit

CONTACTS AND LOCATIONS:
Locations (55):
- United States (55):
  - Urology Centers of Alabama, Homewood, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Arkansas Urology, Little Rock, Arkansas
  - Pacific Clinical Center, Encino, California
  - Los Angeles Clinical Research Center, Encino, California
  - Urology Associates of Central California, Fresno, California
  - Center for Urologic Research, La Mesa, California
  - South Orange County Medical Research Center, Laguna Woods, California
  - San Diego Uro-Research, San Diego, California
  - Western Clinical Research, Torrance, California
  - Urology Research Options, Aurora, Colorado
  - Connecticut Clinical Research Center, Waterbury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Atlantic Urological Associates, Daytona Beach, Florida
  - UroSearch, Inverness, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Atlantic Urological Associates, New Smyrna Beach, Florida
  - UroSearch, Ocala, Florida
  - Florida Foundation for Healthcare Research, Ocala, Florida
  - Atlantic Urological Associates, Orange City, Florida
  - Atlantic Urological Associates, Saint Augustine, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Urology, PA, Atlanta, Georgia
  - West Side Veteran Administration Medical Center, Chicago, Illinois
  - Kankakee Urological Associates, Kankakee, Illinois
  - Specialty Care Research, Peoria, Illinois
  - Welborn Clinic East, Evansville, Indiana
  - Northeast Indiana Research, Fort Wayne, Indiana
  - Urology of Indiana, LLC, Indianapolis, Indiana
  - Urological Associates, PC, Davenport, Iowa
  - 206 Research Associates, Greenbelt, Maryland
  - Lawrenceville Urology, Saint Joseph, Michigan
  - Kansas City Urology Care, Kansas City, Missouri
  - Saint Louis Urological Surgeons, Inc, St Louis, Missouri
  - Sheldon J. Freedman, MD, LTD, Las Vegas, Nevada
  - Nevada Urology Associates, Reno, Nevada
  - Urological Surgical Associates, Edison, New Jersey
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Associated Urologic Specialists, PA, Marlton, New Jersey
  - Suffolk Urology Associates, Bay Shore, New York
  - Urological Surgeons of Long Island, Garden City, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - Center for Urologic Research of Western New York, Williamsville, New York
  - Northeast Urology Research, Concord, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - University Urological Research Institute, Providence, Rhode Island
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Vanderbilt Medical Center Dept of Urologic Surgery, Nashville, Tennessee
  - Urology Specialists & Associates, Dallas, Texas
  - Urology Associates of North Texas, Fort Worth, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - Devine-Tidewater Urology, Virginia Beach, Virginia
  - Madigan Army Medical Center, Tacoma, Washington